CLINICAL TRIAL: NCT06619106
Title: Development of a Cognitive Tool for Rapid and Reliable Screening of Minimal Hepatic Encephalopathy: Pilot Study
Acronym: BLOCK-HE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231310
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Pathology (Fibrosis, Cirrhosis, Porto Systemic Shunts)
Keywords: Hepatic encephalopathy; hepatic failure; neuropsychology; neurology; cognitive tools
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Liver Failure | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Population with chronic liver disease or the presence of portal-systemic shunts, attending the BLIPS day hospital
  Interventions: Other: Cognitive test

INTERVENTIONS:
Other: Cognitive test — Cognitive test based on building blocks

SUMMARY:
The aim of this project is to evaluate the sensitivity and specificity of a cognitive test toward the presence of minimal hepatic encephalopathy (MHE). MHE is a neurological complication due to hepatic dysfunction and/or the presence of porto-systemic shunts defined by the presence of neurocognitive impairments (NI). Other factors of brain injury may cause NI independently from the liver condition making the differential diagnosis difficult using available cognitive tests (ANT Animal Naming Test, PHES Psychometric Hepatic Encephalopathy Score, CFF Critical Flicker Frequency test). The cognitive test evaluated in this project is a construction task using construction blocks, allowing the evaluation of psychomotor speed, executive functions, attention, and episodic memory. The measures will be compared to other cognitive tests validated for the evaluation of the targeted cognitive functions (PHES, Mesulam Cancelling task, Rey-Osterrieth complex figure, Free and Cued Selective Reminding Test) and cognitive tests validated for the diagnosis of MHE (PHES, ANT, CFF). The diagnosis of MHE is based on an adjudication committee including a multimodal assessment of MHE (brain MRI with spectroscopy, EEG, blood sample, neuropsychological assessment), allowing the evaluation of comorbidities such as other factors of brain injury.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE), corresponding to all the neurocognitive symptoms caused by liver damage and/or the presence of portosystemic shunts. HE can take several forms depending on its intensity, ranging from subtle neuropsychological abnormalities that are difficult to detect during a routine interview ("minimal" HE, MHE) to temporospatial disorientation and confusion that can lead to coma ( "overt" HE, OHE). MHE can significantly impair the quality of life of patients and caregivers; it is associated with a poorer prognosis of liver pathology and a significantly more frequent occurrence of OHE. Detection of MHE is complex, and involves the convergence of a large number of tests recognized as sensitive: venous ammonia level, electroencephalogram, MRI with spectroscopy, complete neuropsychological assessment. Today, there is no unanimously recognized Gold Standard.

The objective of this research project is to develop a cognitive test to detect HE sensitively and specifically, in order to detect HE.

To do this, the investigators will evaluate the qualities of a rapid and accessible test. It is a test made up of building blocks to assess psychomotor speed, attention, executive functions and episodic memory. If it proves sensitive and specific enough for the diagnosis of MHE, it could be disseminated and allow the screening of MHE.

To do this, the investigators will compare the block construction test to other neuropsychological examinations validated in the diagnosis of MHE (PHES: Psychometric Hepatic Encephalopathy Score, CFF: Critical Flicker Frequency test, ANT: Animal Naming Test). These examinations are reference cognitive tests in the diagnosis of MHE, but the results between these tests diverge and do not currently make it possible to replace all of the clinical examinations described above. The investigators will also compare the construction block test to cognitive tests validated for the evaluation of the targeted cognitive functions (ROCF Rey-Osterrieth complex figure, FCSRT Free and Cued Selective Reminding test, MCT Mesulam cancelling task). The diagnosis of MHE is based on an adjudication committee including a multimodal assessment of MHE (brain MRI with spectroscopy, EEG, blood sample, neuropsychological assessment), allowing the evaluation of comorbidities such as other factors of brain injury.

Main objective : to evaluate the sensitivity and specificity of the construction test to the presence of MHE.

Secondary objectives:

1. Comparison of screening qualities of the construction test to MHE diagnosis validated tests (PHES, CFF, ANT)
2. Evaluate the impact of the presence of comorbidities (factors of brain injury) in the results of the construction test.
3. Evaluate the psychometric qualities of the construction test compared to validated neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Hepatic pathology (fibrosis, cirrhosis, porto-systemic shunts)
* Evaluation at BLIPS clinic (neuropsychological assessment, MRI, EEG and blood sample with ammonia)

Exclusion Criteria:

* Opposition to participating in the study
* Not being affiliated with French healthcare system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis or portosystemic shunts with suspicion of minimal hepatic encephalopathy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-09-18 (Estimated); Study Completion 2027-09-18 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of the construction test according to the diagnosis of MHE, after construction of a logistic model. | between day 0 and 14 from inclusion

SECONDARY OUTCOMES:
Comparison of the sensitivities and specificities of the construction test compared to the MHE reference tests | Between day 0 and 14 from inclusion
  Comparison of the sensitivities and specificities of the construction test compared to the MHE reference tests like: PHES (Psychometric Hepatic Encephalopathy Score), CFF (Critical Flicker Frequency test), ANT (Animal Naming Test)
Evaluate the sensitivity and specificity of the construction test for the diagnosis of hepatic encephalopathy, taking into account the presence of neurological comorbidities. | Between day 0 and 14 from inclusion
Correlation analysis between subsets of the construction test (planning, speed, selective attention, memory) with reference cognitive tests assessing these cognitive functions | Between day 0 and 14 from inclusion
  Correlation analysis between subsets of the construction test (planning, speed, selective attention, memory) with reference cognitive tests assessing these cognitive functions like: ROCF (Rey-Osterrieth complex figure), FCSRT (Free and Cued Selective Reminding test), MCT (Mesulam cancelling task), PHES subtests (Psychometric Hepatic Encephalopathy Score)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas WEISS, MD,PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Dominique THABUT, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hepato-gastro-enterology department, Pitié Salpêtrière hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.